CLINICAL TRIAL: NCT06767111
Title: Multi-center, Two-arm Clinical Study Evaluating the Performance of the Techcyte Sureview Cervical Cytology System and Its Subsystems for the Assessment of Pap Tests
Brief Title: Techcyte SureView Cervical Cytology System Clinical Validation Study
Status: Enrolling by invitation | Type: Observational
Sponsor: Techcyte, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1-VAL-3427
Record Dates: First submitted 2025-01-06; First posted 2025-01-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-09

CONDITIONS: Cervical Cytology; PAP
Keywords: in vitro diagnostic device; IVD; AI; whole slide scanner; pap test slide; pap; cervical cytology; digital pathology; digital cytopathology

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Pap test slides prepared using the ThinPrep and SurePath methods. These slides are prepared prior to the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | Unapproved Device: Yes | US Export: No

INTERVENTIONS:
Device: Digital cervical cytology slide imaging system with artificial intelligence (AI) algorithm in vitro diagnostic (IVD) device — Digital cervical cytology slide imaging system with artificial intelligence (AI) algorithm to be used for AI-assisted review

SUMMARY:
The clinical study is a multi-center, retrospective, blinded, matched-pair, two-arm clinical study in which one test assessment and a control assessment of liquid-based cytology (LBC) pap tests are performed and compared to a reference.

The control method is defined as the assessment of LBC pap tests performed by a cytotechnologist (CT) and/or cytopathologist (CP) using standard laboratory cervical cytology practices (i.e. a manual assessment) and following The Bethesda System for Reporting Cervical Cytology (TBS). The control method is referred to as the "standard method".

The test method is referred to as the AI-assisted method. The AI-assisted method is defined as the assessment of the same LBC pap test as in the standard method, but with the Techcyte SureView Cervical Cytology System, which has pap tests being scanned on the Pramana SpectralHT Cubiq whole slide scanner, analyzed with the Techcyte Cervical Cytology Algorithm (TCCA) and presented on the Techcyte Viewer, using the Dell U3223QE Monitor for assessment by a CT/CP following the TBS.

In addition, the time spent reviewing the samples with both methods will be measured such that the CT workload limit for AI-assisted assessment can be established.

The LBC pap tests to be assessed in the clinical study must have been prepared with either ThinPrep® Pap Test (Hologic) or BD SurePath™ (Beckton, Dickinson and Company). The study aims to enroll for each preparation method an equal number of samples.

ELIGIBILITY:
Inclusion Criteria:

* Glass slides with cervical cytology specimens prepared with Hologic ThinPrep according to the pap test manufacturers Instructions for Use (IFU) using any of Hologic's processors (i.e. ThinPrep2000, ThinPrep 3000, ThinPrep 5000, ThinPrep Genesis). OR Glass slides with cervical cytology specimens prepared with BD SurePath according to the pap test manufacturers IFU using any of BD's processors (i.e. BD Totalys MultiProcessor, BD Totalys SlidePrep, BD PrepStain).
* Slide has the original diagnosis available.
* Slides that fit within the required sample size strata using the sample collection procedure.
* Glass slides with QR code, barcodes, or plain text labels.
* Glass slides with coverslips.
* Slides that are 5 years old or less, except where rare specimens require it. Those specimens will have to be reviewed for degradation per the sample collection procedure.
* Only one sample per patient and all are to be collected, processed and scanned.

Exclusion Criteria:

* Broken or cracked slides.
* Slides with air bubbles or scratched, cracked or broken/missing cover slips.
* Slides with markings (e.g., handwritten pen marking) that cannot be removed according to standard laboratory procedures.
* Degraded slides (ex: slides whose stains have lost color or specimens that are not intact).
* Glass slides with cervical cytology specimens prepared with methods other than Hologic ThinPrep or BD SurePath.
* Glass slides with specimens other than cervical cytology specimens.
* Slides from the same patient.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Samples collected in the United States
Sampling Method: Probability Sample
Enrollment: 4596 (Estimated)
Dates: Start 2024-12-01 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Sensitivity and specificity when comparing pap tests using the Techcyte SureView Cervical Cytology System | 1 day
  The primary objective of the study is to show that the assessment of LBC pap tests using the Techcyte SureView Cervical Cytology System, i.e. the AI-assisted method, is non-inferior to current standard practice, i.e., the standard method, at the LSIL+ threshold used for cytologic diagnosis (specimen adequacy and descriptive diagnosis) as defined by The Bethesda System for Reporting Cervical Cytology.

CONTACTS AND LOCATIONS:
Locations (1):
- Techcyte, Orem, Utah, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Nayar R, Wilbur DC. (eds), The Bethesda System for Reporting Cervical Cytology: Definitions, Criteria, and Explanatory Notes. 3rd ed. Cham, Switzerland: Springer: 2015.